CLINICAL TRIAL: NCT00000379
Title: Treatment of Outcomes of Fluoxetine vs EMDR in PTSD
Brief Title: Fluoxetine vs EMDR to Treat Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01MH058363 (NIH); R01MH058363 (NIH); DSIR AT-CT
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Adult; Comparative Study; Desensitization, Psychologic; Eye Movements; Female; Fluoxetine; Human; Male; Placebos; Stress Disorders, Post-Traumatic; Treatment Outcome; Desensitization, Psychologic -- *methods; Fluoxetine -- *therapeutic use; Stress Disorders, Post-Traumatic -- *therapy; Stress Disorders, Post-Traumatic -- drug therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic | interventions — Fluoxetine; Eye Movement Desensitization Reprocessing

INTERVENTIONS:
Drug: Fluoxetine
Behavioral: EMDR

SUMMARY:
The purpose of this study is to compare two treatments for post-traumatic stress disorder (PTSD): fluoxetine (an antidepressant) and Eye Movement Desensitization and Reprocessing (EMDR, a psychological treatment in which the patient is led through the memory of a traumatic experience in order to heal him/herself).

There are a variety of therapies used to treat PTSD, but the effectiveness of medication alone vs an exposure treatment, such as EMDR, has not been tested.

Patients will be assigned randomly (like tossing a coin) to one of three groups for 8 weeks of treatment. Group 1 will receive fluoxetine; Group 2 will receive EMDR; and Group 3 will receive inactive placebo. Patients will then stop treatment and have evaluations, including psychological tests, at the time treatment is stopped, 8 weeks later, and at 6 months.

An individual may be eligible for this study if he/she:

Has PTSD and is 18 to 65 years old.

DETAILED DESCRIPTION:
To compare the short-term and long-term efficacy of two different treatment approaches in widespread use in clinical settings for treating patients with post-traumatic stress disorder (PTSD): fluoxetine (which acts directly on biological systems) vs a psychological treatment, Eye Movement Desensitization and Reprocessing (EMDR). To clarify: 1) the differential treatment effects of these different treatment modalities; 2) whether symptom improvement is accompanied by changes in pathophysiology; and 3) the long-term effectiveness of these treatments.

In recent years a variety of treatment approaches have been shown to be effective in the treatment of PTSD. These include prolonged exposure therapies (PE), stress inoculation training (SIT), EMDR and psychopharmacological treatment with serotonin re-uptake blockers. While PE has been compared with SIT and a study is currently under way comparing cognitive-behavioral treatment with EMDR, no study as yet has compared the relative merits of pharmacotherapy alone vs an exposure treatment. While it is commonly held that, in order to recover, people with PTSD need to "process" their traumatic memories, treatments that do not involve the processing of traumatic memories (such as SIT or pharmacotherapy) may be just as effective. In clinical practice, many patients with PTSD appear to be effectively treated with pharmacological agents alone, without trauma-focused therapy.

Patients are randomly assigned to one of three conditions: 1) a double-blind psychopharmacological treatment (fluoxetine); 2) a manualized treatment which focuses on "processing" traumatic memories (EMDR); or 3) a placebo control group. After 8 weeks of active treatment, subjects are evaluated, cease treatment, and are assessed again after another 8 weeks and at 6 months in order to evaluate the long-term effects. Training raters remain blind to the subjects' treatment condition throughout the study. Treatment outcome is assessed with a multi-modal psychological and biological assessment battery including: 1) standard psychological tests for PTSD (CAPS); 2) neuroendocrine function (cortisol); and 3) psychophysiological response to traumatic scripts (pre-post changes in heart social and occupational functioning). Treatment adherence is monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Post-Traumatic Stress Disorder (PTSD).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Bessel Van Der Kolk, MD, Principal Investigator
Locations (1):
- The Trauma Center, Brookline, Massachusetts, United States